CLINICAL TRIAL: NCT02058719
Title: Immunosuppressive Effects of Smoking and HIV-1 on the Development of Lung Disease.
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2986
Record Dates: First submitted 2014-02-05; First posted 2014-02-10 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: HIV; Smoking; COPD
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and bronchoscopy (BAL) samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Cohort A1: HIV positive smokers
- Cohort A2: HIV positive non-smokers
- Cohort A3: HIV negative smokers
- Cohort A4: HIV negative non-smokers
- Cohort B1: HIV positive with COPD
- Cohort B2: HIV positive without COPD (non-COPD)
- Cohort B3: HIV negative with COPD

SUMMARY:
This study plans to learn more about pulmonary complications of human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS). Even though antiretroviral therapy (ART) has dramatically decreased the number of opportunistic infections and deaths in HIV infected patients, pulmonary complications (including chronic obstructive pulmonary disease (COPD) development and pneumonias resulting in decreased lung function) of HIV/AIDS continue to be a major cause of morbidity and mortality in this population. The mechanisms underlying the increased risk of COPD and decreased lung function in HIV infected individuals is not well understand and needs to be studied.

The investigators hypothesize that the immunoregulatory consequences and immunosuppressive lung milieu secondary to HIV and cigarette smoke combine to increase the risk of lung infection and injury in HIV infected smokers, hastening the development of COPD. The mechanisms will be directly tested using blood and bronchial alveolar lavage (BAL) cells from smokers and nonsmokers with and without HIV infection.

DETAILED DESCRIPTION:
The first component of this study will be a longitudinal, prospective, 24 weeks study of the effects of HIV-1 infection on innate and acquired immunity in the lung (Cohort A). The second component of this study will be a cross-sectional, case-control study of lung function and immune dysregulation of HIV-1 infected persons on long-term ART (Cohort B).

Cohort A will consist of 120 subjects, stratified by HIV-1 and smoking status

Cohort B will consist of 90 subjects stratified by chronic obstructive pulmonary disease (COPD) and HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria (Cohort A):

* Subjects with chronic HIV-1 infection (Cohorts A1 and A2)
* ART naïve or off all ART for >6 months (Cohorts A1 and A2)
* HIV-1 RNA level >1,000 copies/ml (Cohorts A1 and A2)
* HIV-1 seronegative with no high-risk exposure in the past 30 days (Cohorts A3 and A4)
* 18 years and older (All Cohort A)
* Active cigarette smoker (Cohorts A1 and A3)

Inclusion Criteria (Cohort B):

* Age from 30 to 70 years
* Subjects with chronic HIV-1 infection (Cohorts B1 and B2)
* Subjects on stable 3-drug ART regimen with plasma HIV-1 RNA <50 copies/mL for past 6 months (Cohorts B1 and B2)
* HIV-1 seronegative with no high-risk exposure in the past 30 days (Cohort B3) COPD: forced expiratory volume at one second (FEV1)/forced vital capacity (FVC) <70% and forced expiratory volume (FEV), 45-100% of predicted (Cohort B1 and B3)
* Non-COPD: FEV/FVC >70% and an FEV, >80% of predicted (Cohort B2)

Exclusion Criteria (Cohort A and B):

* Pregnancy
* Weight less than 110 pounds (for venipuncture)
* Patient inability to participate in the study and undergo venipuncture and bronchoscopy procedures
* Use of systemic or inhaled corticosteroids in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive (smokers and non-smokers) and negative subjects (smokers and non-smokers) will be recruited. HIV positive (with and without COPD) and HIV negative with COPD will also be recruited. All subjects will be between ages 18 and 70.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The change in immunoregulatory markers: PD-1 expression and interleukin (IL)-10 production by alveolar macrophages (AMs) from baseline to week 24. | Baseline, Week 24
  Evaluate the immunoregulatory change between HIV positive (smokers/non-smokers) and HIV negative (smokers/non-smokers)
PD-1 expression and IL-10 production by AMs at baseline | Baseline
  Evaluate the association of PD-1 expression and IL-10 production by AMs after long-term antiretroviral therapy (ART) with abnormal lung function and a COPD phenotype between HIV positive (with and without COPD) and HIV negative with COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B. Campbell, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States